CLINICAL TRIAL: NCT01814059
Title: A Phase 1, Open-Label Study of Sirolimus in Eosinophil-Associated Gastrointestinal Disorders
Brief Title: Sirolimus for Eosinophil-Associated Gastrointestinal Disorders
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130094; 13-I-0094
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-05-12

CONDITIONS: Eosinophilic Gastroenteritis; Eosinophilic Esophagitis
Keywords: Sirolimus; Eosinophilic Esophagitis; Eosinophilic Gastroenteritis; T -Cells; Food Allergy
MeSH Terms: conditions — Eosinophilic enteropathy; Eosinophilic Esophagitis; Food Hypersensitivity | interventions — Sirolimus

INTERVENTIONS:
Drug: sirolimus

SUMMARY:
Background:

* Eosinophil-associated gastrointestinal disorders (EGID) are a group of related disorders that affect the esophagus, stomach, and bowel. There are two major types of EGID, eosinophilic esophagitis and eosinophilic gastroenteritis. They are caused by the body's immune system being activated by food allergens, which then damages the gut wall. People with EGID have large numbers of eosinophils (a type of white blood cell) in their gut. EGID can cause difficulty swallowing, abdominal pain, or nausea.
* At present, there are no drugs specifically approved to treat EGID. Most adults who have EGID receive steroid therapy to manage the symptoms. However, long-term steroid use may cause other problems in the body. Researchers want to see if low-dose sirolimus can be used to treat EGID. Sirolimus is a drug used to prevent rejection of transplanted organs. It may be able to keep the body's immune cells from being activated by food allergens and decrease the eosinophils.

Objectives:

- To see if low dose sirolimus is safe and decreases blood or gut eosinophils in EGID.

Eligibility:

* Individuals between 18 to 65 years of age who have EGID.
* Participants must also have an elevated blood eosinophil count and positive blood tests for IgE antibodies to foods.

Design:

* Participants who are on medicine for EGID or related symptoms must be on a stable dose for 1 month before screening and stay on that dose throughout the study.
* Participants will be screened with a medical history and physical exam, and review their symptoms. They will provide blood and urine samples. They will also have heart and lung function tests. Some participants may have allergy skin tests.
* At the first study visit, participants will have 2 days of inpatient tests. They will repeat the tests from the screening visit. They will also have a full analysis of the esophagus, stomach, and small intestine. On the second day, they will start to take sirolimus as a liquid with orange juice or water.
* Participants will continue to take sirolimus at home. They will record their doses and any symptoms. They will also have a visit to provide blood samples about 2 weeks after the first study visit.
* At the second study visit (about a month after the first visit), participants will repeat the tests from the screening visit. The sirolimus dose may be adjusted as needed.
* Participants will take sirolimus for at least another 28 days. Depending on the dose of the drug and the blood test results, some participants may need to take it for up to 112 days. Those who take the drug for a longer period will have additional study visits with tests.
* There will be another study visit when participants stop taking the drug. The last visit will be a final follow-up visit.

DETAILED DESCRIPTION:
Eosinophil-Associated Gastrointestinal Disorders (EGID) are a group of related disorders characterized by gastrointestinal symptoms and eosinophilic infiltration of the gastrointestinal wall. The 2 major forms of EGID, eosinophilic esophagitis (EoE) and eosinophilic gastroenteritis (EG), differ in regard to the site of inflammation (esophagus vs. stomach/small bowel). Both EoE and EG are highly associated with coexisting allergic disease, and a large fraction of EGID patients are sensitized to multiple food allergens. Existing data strongly support the concept that EGID is a food-allergen-driven, eosinophilic, inflammatory gut disease. Multiple lines of evidence support a major role for Th2 cells and the cytokines they express (IL-4, IL-5, and IL-13) in EGID pathogenesis.

There are presently no drugs with a labeled indication for EGID. Most adult patients are managed long-term with corticosteroid therapy, which raises concerns about toxicity. Sirolimus is an immunomodulator approved for use in preventing transplant rejection. It specifically inhibits Th2 cell proliferation in vitro, suggesting it may have activity in EGID.

This study is a phase I open-label design intending to target a sirolimus whole blood concentration of 6 ng/mL for a duration of 56 days. Twenty adult EGID subjects 10 with EoE and 10 with EG with evidence of Th2-mediated IgE sensitization and peripheral blood eosinophil counts (Bullet)800 cells/ L will be recruited to participate. Subjects will begin sirolimus at a dose of 1.2 mg/m2/day. Blood sirolimus level will be checked at 14- to 28-day intervals, and the dose will be serially adjusted in each subject as needed to target the 6- ng/mL target trough concentration. Blood will be drawn at each visit to monitor drug levels and safety labs.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals will be eligible for study participation if they meet all of the following criteria:

1. Age greater than or equal to18 years and less than or equal to 65 years at the time of Study Visit 1.
2. Presence of the following diagnostic criteria for EGID:

   1. Subjects with EoE must have: 1) esophageal symptoms; 2) histologic evidence of esophageal tissue infiltration by eosinophils with a peak greater than or equal to25 eosinophils per high-powered field (while on greater than or equal to 2 months of twice daily proton-pump inhibitor therapy); and 3) no known etiology for the tissue eosinophilia despite careful clinical evaluation.
   2. Subjects with EG must have: 1) gastrointestinal symptoms; 2) histologic evidence of stomach or duodenal tissue infiltration by eosinophils with a peak greater than or equal to35 eosinophils per high-powered field; and 3) no known etiology for the tissue eosinophilia despite careful clinical evaluation.
3. Blood AEC greater than or equal to 800 cells/microL at the screening visit. This screening value will not be used to calculate the baseline AEC used in the principal secondary endpoint.
4. Baseline laboratory values within the following ranges:

   1. White blood cell count greater than or equal to3,300 cells/microL.
   2. Absolute neutrophil count greater than or equal to1,000 cells/microL.
   3. Hemoglobin greater than or equal to10 g/dL.
   4. Platelet count greater than or equal to100,000 platelets/microL.
5. Three or more positive allergen-specific IgE tests (skin tests or in vitro assay) out of this panel of 10 food and aeroallergens: milk, eggs, wheat, soy, shrimp, cod, corn, peanut, dust mite, cat.
6. Subjects currently on medication for their EGID or for GI symptoms must be on a stable dose for 1 month prior to screening and be willing to continue on that dose for the duration of the study. Other medications (e.g. for hypertension, asthma, or depression) may be adjusted by the subject s physician.
7. Willingness to have samples stored for future research and genetic testing.
8. Women of childbearing potential must have a negative serum beta-hCG.
9. Agree to practice abstinence or effective contraception as detailed below.

Contraception: The fetal risks associated with sirolimus are not known, but pre-clinical animal data demonstrate some risk. Subjects must agree not to become pregnant or impregnate a female, accordingly. Females of childbearing potential must have a pregnancy test at each NIH visit. Because of the risk involved, both male and female subjects and their partners must use 2 methods of birth control. As per the sirolimus package insert, subjects must continue to use both methods for 3 months after stopping the study drug. Two methods of birth control may be selected from the list included below:

* Hormonal contraception.
* Male or female condoms with or without a spermicidal.
* Diaphragm or cervical cap with a spermicidal.
* Intrauterine device.

If pregnancy is suspected or should occur, subjects must notify the study staff immediately.

EXCLUSION CRITERIA:

Individuals will not be eligible to participate in this study if they meet any of the following criteria:

1. Are breast feeding.
2. Are HIV positive or have any other known immunodeficiency.
3. Have used any investigational agent within 6 months of the screening visit.
4. Express the FIP1L1-PDGF-R fusion gene.
5. Have evidence of preexisting proteinuria with urine albumin-to-creatinine ratio >200 mg/g (men) or >300 mg/g (women).
6. Have serum creatinine with estimated GFR <60 mL/min/1.73 m2.
7. Have any chronic liver disease, including hepatitis B or C.
8. Use of medications that have CYP3A4 or P-glycoprotein (P-gp) inhibitor or inducer activity.
9. Are Taking ACE inhibitor medicatons
10. Drug allergy or intolerance to allergies to sirolimus, other rapalogs, or excipients in the preparation.
11. Have any condition that, as determined by the investigator, places the patient at undue risk by participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-03-07; Primary Completion 2015-05-12 (Actual); Study Completion 2015-05-12 (Actual)

PRIMARY OUTCOMES:
Assess safety of sirolimus in patients with eosinophilic gastrointestinal disorders. | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Calman P Prussin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Straumann A, Conus S, Grzonka P, Kita H, Kephart G, Bussmann C, Beglinger C, Smith DA, Patel J, Byrne M, Simon HU. Anti-interleukin-5 antibody treatment (mepolizumab) in active eosinophilic oesophagitis: a randomised, placebo-controlled, double-blind trial. Gut. 2010 Jan;59(1):21-30. doi: 10.1136/gut.2009.178558. PMID 19828470
- [Background] Jyonouchi S, Brown-Whitehorn TA, Spergel JM. Association of eosinophilic gastrointestinal disorders with other atopic disorders. Immunol Allergy Clin North Am. 2009 Feb;29(1):85-97, x. doi: 10.1016/j.iac.2008.09.008. PMID 19141344
- [Background] Stein ML, Collins MH, Villanueva JM, Kushner JP, Putnam PE, Buckmeier BK, Filipovich AH, Assa'ad AH, Rothenberg ME. Anti-IL-5 (mepolizumab) therapy for eosinophilic esophagitis. J Allergy Clin Immunol. 2006 Dec;118(6):1312-9. doi: 10.1016/j.jaci.2006.09.007. Epub 2006 Nov 7. PMID 17157662